CLINICAL TRIAL: NCT06364319
Title: Study on the Efficacy and Safety of Anti-CD25 rhMAb in the Treatment of Steroid-Refractory Chronic Graft-Versus-Host Disease (cGVHD) of the Liver Following Allogeneic Hematopoietic Stem Cell Transplantatio
Brief Title: Efficacy and Safety of Anti-CD25 rhMAb in the Treatment of Steroid-Refractory cGVHD
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Director, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024PHD002-001
Record Dates: First submitted 2024-03-20; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: cGVHD
MeSH Terms: interventions — Prednisone; ruxolitinib; Cyclosporine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti-CD25 rhMAb + traditional therapy (Experimental)
  Interventions: Drug: anti-CD25 rhMAb; Drug: Prednisone; Drug: Ruxolitinib; Drug: Cyclosporine
- traditional therapy (Placebo Comparator)
  Interventions: Drug: Prednisone; Drug: Ruxolitinib; Drug: Cyclosporine

INTERVENTIONS:
Drug: anti-CD25 rhMAb — 1 mg/kg/day administered IV day 1, 4, and 8, then weekly for 6 doses. For patients achieving partial remission, an extra dose of Anti-CD25 rhMAb can be given on days 39 and 49.
  Arms: Anti-CD25 rhMAb + traditional therapy
Drug: Prednisone — Maintain pre-screening dose
Drug: Ruxolitinib — 10mg, BID PO
Drug: Cyclosporine — 1.25mg/kg, BID PO/IV, target:150-250ng/ml

SUMMARY:
The study plan aims to include patients who have been diagnosed with steroid-refractory chronic GVHD in the liver following allogeneic hematopoietic stem cell transplantation. After obtaining informed consent, the patients will be randomly assigned to either the Anti-CD25 rhMAb treatment group or the traditional treatment group. The objective is to assess the effectiveness and safety of Anti-CD25 rhMAb in the treatment of severe chronic GVHD affecting the liver.

ELIGIBILITY:
Inclusion Criteria:

1. Age 16 and 65 years
2. Received allogeneic hematopoietic stem cell transplantation
3. Developed chronic GVHD in the liver after transplantation
4. Ineffective prednisone treatment prior to screening
5. Received ≤4 lines of systemic therapy prior to screening
6. After informed consent, the patient agreed to receive anti-CD25 rhMAb treatment

Exclusion Criteria:

1. Elevation of bilirubin, ALT, or alkaline phosphatase due to reasons other than chronic GVHD
2. No prior treatment with prednisone
3. Overlap syndrome
4. Uncontrolled active infection
5. Organ failure
6. Early progression or recurrence of hematologic diseases
7. Allergy to anti-CD25 rhMAb
8. Received other interleukin-2 receptor monoclonal antibody treatment due to various reasons within one month after transplantation
9. Participated in other clinical studies within one month

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
overall response rate (ORR) | 56 days
  ORR is defined as the percentage of complete response (CR) and partial response (PR).

SECONDARY OUTCOMES:
duration of response（DOR） | 1 year
  DOR is defined as the duration calculated from the time of achieving PR or CR until the progression of GVHD, the addition of other systemic immunosuppressive therapy, or death.
patient-reported outcomes (PRO) | 1 year
  Based on the Lee Chronic GVHD Symptom Scale.
disease-free survival (DFS) | 1 year
  DFS is defined as the duration of survival after treatment in which the original hematologic disease is in a state of complete remission.
failure-free survival (FFS) | 1 year
  Events that are considered as failures include the onset of new chronic GVHD, relapse, and death.
non-relapse mortality (NRM) | 1 year
  NRM is defined as death due to reasons other than progression/relapse of hematologic disease.
overall survival （OS） | 1 year
  OS is defined as the time from treatment until death from any cause or the last follow-up.
adverse drug reactions (ADR) | 1 year
  The occurrence of various organ toxicities related to treatment that emerge following treatment.

IPD SHARING:
Plan to Share IPD: Undecided
Our plan is to disseminate the findings of this trial via peer-reviewed articles.